CLINICAL TRIAL: NCT06554106
Title: Effects of Neuromuscular Electrical Stimulation in Fibromyalgia Patients
Brief Title: Neuromuscular Electrical Stimulation in Fibromyalgia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Songül Bağlan Yentür, Firat University, Firat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/10-01
Record Dates: First submitted 2024-08-13; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Neuromuscular Electrical Stimulation; Pain
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuromuscular Electrical Stimulation Group (Experimental): All patients will be taught neck normal joint movement exercises, upper trapezius stretching exercise and posture exercises. In addition to the study group, NMES will be applied to the upper trapezius muscle for 30 minutes 5 days a week for 4 weeks. Neuromuscular Electrical Stimulation (NMES) applications will be performed with a Compex 3 (Compex Medical SA, Ecublens, Switzerland) model, portable and programmable electrostimulator unit in rehabilitation mode and under the supervision of an expert physiotherapist experienced in the device and application. The NMES program will be applied with a 4-channel device with a functional stimulation capacity of 120 mA, pulse duration 400 μs and pulse frequency 150 Hz.
  Interventions: Other: Neuromuscular Electrical Stimulation Group
- Control group (Experimental): Patients will be taught neck normal joint movement exercises, upper trapezius stretching exercise and posture exercises.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Neuromuscular Electrical Stimulation Group — All patients will be taught neck normal joint movement exercises, upper trapezius stretching exercise and posture exercises. In addition to the study group, NMES will be applied to the upper trapezius muscle for 30 minutes 5 days a week for 4 weeks. Neuromuscular Electrical Stimulation (NMES) applications will be performed with a Compex 3 (Compex Medical SA, Ecublens, Switzerland) model, portable and programmable electrostimulator unit in rehabilitation mode and under the supervision of an expert physiotherapist experienced in the device and application. The NMES program will be applied with a 4-channel device with a functional stimulation capacity of 120 mA, pulse duration 400 μs and pulse frequency 150 Hz.
  Arms: Neuromuscular Electrical Stimulation Group
Other: Control Group — Patients will be taught neck normal joint movement exercises, upper trapezius stretching exercise and posture exercises.
  Arms: Control group

SUMMARY:
Fibromyalgia syndrome (FMS) is associated with chronic widespread pain and at least eleven positive tender points out of 18 according to the American College of Rheumatology (ACR) 1990 criteria. Neuromuscular electrical stimulation (NMES) stimulates nerve fibers providing innervation in healthy muscle and muscle fibers in denervated muscle to produce contraction. All patients will be taught neck normal joint motion exercises, upper trapezius stretching exercise and posture exercises. Patients included in the study will be randomly distributed equally between the two groups. In addition to the study group, NMES will be applied to the upper trapezius muscle for 30 minutes 5 days a week for 4 weeks. Pain, disability and sleep quality of all patients will be evaluated.

DETAILED DESCRIPTION:
Fibromyalgia syndrome (FMS) is associated with chronic widespread pain and at least eleven positive tender points out of 18 according to the 1990 criteria of the American College of Rheumatology (ACR) (1). Pain and other symptoms associated with fibromyalgia interfere with daily functions, work and social activities, leading to a decrease in quality of life. Neuromuscular electrical stimulation (NMES) stimulates nerve fibers that provide innervation in healthy muscle and muscle fibers in denervated muscle to produce contraction. Studies on TENS current in patients with FM have shown that pain decreases and functional status improves. However, although muscle weakness has been described in patients with FM, there are no studies on the effects of NMES application. All patients will be taught neck normal joint motion exercises, upper trapezius stretching exercise and posture exercises. Patients included in the study will be randomly distributed equally between the two groups. In addition to the study group, NMES will be applied to the upper trapezius muscle for 30 minutes 5 days a week for 4 weeks. Pain, disability and sleep quality of all patients will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were aged between 18-65 years,
* Patients who got diagnosed with Fibromyalgia Syndrome

Exclusion Criteria:

* Patients who had regular exercise habits, malignancy, pregnancy, incorporation
* Patients who had changes of medical treatment in last 3 months
* Patients who had dysfunction that can prevent physical activity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-20 (Estimated); Primary Completion 2024-10-20 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Pain assessment | 1 minute
  Pain intensity will be evaluated according to VAS. Patients will be asked to mark the pain intensity on a 10 cm line. 0 means no pain and 10 means unbearable pain.

SECONDARY OUTCOMES:
Disability assessment | 2 minutes
  Fibromyalgia Impact Questionnaire will be used. The FIQ consists of 10 items. The first item includes daily activity questions scored on a Likert scale from 0 to 3 (always able to do - never able to do).
Sleep quality assessment | 2 minutes
  Pittsburg Sleep Quality Index will be used to evaluate sleep quality

CONTACTS AND LOCATIONS:
Locations (1):
- Songul Baglan Yentur, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No